CLINICAL TRIAL: NCT02230267
Title: High-intensity Exercise and Fall Prevention Boot Camp for Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nevada, Las Vegas (Other)
Responsible Party: Principal Investigator, Merrill Landers, Chair and Associate Professor, University of Nevada, Las Vegas
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTR-IN UNLVPT 2014.01
Record Dates: First submitted 2014-08-27; First posted 2014-09-03 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Parkinson's Disease
Keywords: boot camp; exercise; balance training; fall prevention; falling; strength training
MeSH Terms: conditions — Parkinson Disease; Motor Activity | interventions — Fumigant 93; RE1-silencing transcription factor; Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High intensity boot camp (Experimental): Each of the two HIBCs will have 10 participants (20 total) with a 1:5 physical therapist-to-patient ratio. Each HIBC session will last 1.5 hours and will be held on 4 days of the week. Participants will be required to attend 3 of those 4 days but may attend all. Because this is a pragmatic trial, therapists will have some leeway to control the intensity and the modality of the exercise. However, the basic format of the HIBC will consist of the following exercise components: A. 30 minutes of moderate-high intensity aerobic exercise at 70%+ of estimated maximum heart rate; B. 15 minutes of strengthening the major muscle groups of the trunk and upper/lower extremities; C. 15 minutes of balance training; and, D. 15 minutes of rest and stretching. Participants will rotate through these four different exercise components in a circuit fashion.
  Interventions: Other: High intensity exercise and balance training
- Usual care arm (Active Comparator): The low intensity exercise group will participate in the Fitness Counts Exercise Program (FCEP) which is a basic low intensity, sitting and standing exercise program (10 minutes of stretching, 10 minutes of aerobic exercise (60% of heart rate maximum), and 10 minutes of strengthening). This exercise program was developed by the National Parkinson Foundation and is commonly used in PD exercise classes. The physical therapist-to-patient ratio will be 1:5. As there are two clinical sites, there will be 10 participants in each of the two boot camps (20 total). The FCEP will be 1 hour daily on four days of the week. Participants will be required to attend 3 days per week but may attend more if they are able.
  Interventions: Other: Usual care arm exercise

INTERVENTIONS:
Other: High intensity exercise and balance training
  Other Names: A. 30 minutes of moderate-high intensity aerobic exercise at 70%+ of estimated maximum heart rate; B. 15 minutes of strengthening the major muscle groups of the trunk and upper/lower extremities; C. 15 minutes of balance training; D. 15 minutes of rest and stretching
  Arms: High intensity boot camp
Other: Usual care arm exercise
  Other Names: 10 minutes of stretching; 10 minutes of aerobic exercise (60% of heart rate maximum); 10 minutes of strengthening
  Arms: Usual care arm

SUMMARY:
Several animal and human epidemiologic studies have provided evidence that exercise may be neuroprotective in Parkinson's disease (PD). Exercise may forestall diagnosis and, in the case of those who have already been diagnosed with PD, it may slow the observed neurodegeneration. Unfortunately, because this line of research is in early stages, there is little evidence to indicate what biological mechanisms underlie the neuroprotection that is conferred with exercise. Toward this end, it is possible that an interaction between endogenous antioxidant enzymes, inflammatory processes, and reactive oxygen species may be associated with exercise improvements in PD.

One of the most common reasons for premature death in PD is falls. Several meta-analyses have concluded that exercise training programs focused on balance and/or strength training are effective at improving aspects of balance. Taken together, the current body of evidence suggests that exercise may be neuroprotective and balance/strength training may decrease the likelihood of a fall. The combination of these efficacious treatment modalities (exercise and balance/strength training) in a comprehensive treatment approach to improve PD symptoms and balance has been previously reported at relatively mild or moderate exercise intensities. Because recent research has suggested that patients with PD may benefit more from more physically intense programs, we are proposing a more aggressive approach with regard to exercise intensity and frequency in the present trial. The primary purpose of this study is to determine the feasibility and safety of a high intensity exercise approach to PD. A secondary purpose is to determine the trajectory of change in outcomes over the duration of the trial from a high intensity fall prevention program. It is hoped that a signal of efficacy will allow this trial to progress to a comparative effectiveness trial. An important innovative design element is collecting biological assays to better understand the mechanism underlying the anticipated clinical improvements.

Aim 1 is to test the feasibility of a high-intensity exercise and fall prevention boot camp (HIBC) in patients with PD by analyzing adherence and whether they achieve minimum Centers for Disease Control exercise standards (150 min/wk moderate level aerobic exercise; strengthening at least two times per week) for the duration of the trial. Aim 2 is to determine if participation in an 8-week HIBC under the direction of a physical therapist is safe for individuals with PD. Secondary Aim 3 is to determine if participation in an 8-week HIBC will produce a signal of efficacy for several physical outcomes: falls per physical activity ratio, balance efficacy, motor activity, fatigue, muscle strength, bone health, cognition/mood, and quality of life. Secondary Aim 4 is to determine if participation in an 8-week HIBC will produce a signal of efficacy for biological outcomes, anti-inflammatory cytokines and anti-oxidant enzymes. An additional exploratory aim will be an analysis of BDNF val66val, val66met, met66met polymorphisms to determine if there is a differential response to exercise.

This trial is innovative because it utilizes a high intensity comprehensive exercise treatment approach (aerobic exercise, strengthening, and balance training). To our knowledge, there have been no trials of individuals with PD who have participated in a trial of this intensity in a group "boot camp" setting. Another innovative design element is the use of three novel assessments: biological assays of pro- and anti-inflammatory cytokines, endogenous anti-oxidant enzymes and a novel assessment of falls (falls per physical activity ratio).

Participants will be randomly assigned into either an 8-week HIBC group or an 8-week usual care control group (standard, low intensity group therapy class) under the direction of physical therapists. Each group will have 15 participants with a 1:5 patient-to-therapist ratio. The HIBC will be 1.5 hours daily, Monday through Friday. Participants will be required to attend 3 out of the 5 days. The protocol of the HIBC will include the following exercise components: A. 30 minutes of moderate-high intensity aerobic exercise; B. 15 minutes of strengthening the major muscle groups; C. 15 minutes of balance training; and, D. 15 minutes of interspersed rest and stretching. Participants will rotate through these four exercise components. Participants will have one baseline test and assessments at the 2-week, 4 week, 8-week, and 6-month points. Outcomes of the primary aims (Aim 1 and Aim 2) will be frequency counts of participation, adverse events, and compliance with exercise. The outcomes for the secondary aims will include measures of balance and falls, physical capacity, fatigue, exercise/physical activity behavior, and biological assays.

ELIGIBILITY:
Inclusion Criteria:

* Neurologist-diagnosed idiopathic PD based on the UK PD brain bank criteria
* Aged 45-85
* Hoehn and Yahr stages 1-3 (mild to moderate PD)
* Participants do not anticipate a change in medication or surgical procedures in the next 8 months of the trial (2 months for the trial and 6 for the follow-up)
* Clearance from primary care physician to participate in the trial
* Must be stable on PD medication and DBS for 3 months prior to trial

Exclusion Criteria:

* Poorly controlled or unstable cardiovascular disease that precludes participation in exercise
* Moderate-to-severe dementia using the Montreal Cognitive Assessment (MoCA). We will exclude participants with a MoCA cut off score of <26/30. This cut off value has excellent sensitivity (90%) and specificity (75%).
* Inability to stand or walk for more than 10 minutes
* Other significant disorders that would limit endurance exercise participation (i.e., osteoarthritis, stroke, respiratory problems, traumatic brain injury, neuromuscular disease, pain)
* Already participating in a regular, vigorous exercise program (3X/week or more of >60% estimated maximum heart rate)
* Participants will be excluded from the trial if they are taking any medications that interfere with heart rate response to exercise

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-08; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Frequency feasibility | After completion of the 8 week trial
  The number of participants that attend and participate in the treatment at least 3 times per week for 8 weeks.
Aerobic feasibility | At the end of the 8 week trial
  The number of participants that complete at least 150 minutes per week of moderate intensity exercise (70%+ of their estimated HR maximum). This will be ascertained using heart rate monitors.
Strength feasibility | At the end of the 8 week trial
  The number of participants that participate in strengthening exercises that incorporates all the major muscle groups at least two days per week.
Compliance | At the end of the 8 week trial
  Drop-out rate and reason for drop-out will be tracked.
Safety | Ongoing throughout the 8 week trial
  Exercise-related adverse events (e.g., strains/sprains, cardiovascular events).
Motivation | At 8 weeks
  The Intrinsic Motivation Inventory (IMI) will be used to gather information about motivation.
Falls | At the end of the 8 week trial
  Falls and fall injuries in and out of boot camp will be collected.

SECONDARY OUTCOMES:
Falls | up to 6 months
  Falls will be tracked for 6 months after the boot camp using a falls diary. A member of the research team will call each month to interview participants about their falls. We will assess falls/fall injuries per physical activity ratio during the 6 month period following the trial and time to a fall/fall injury after the trial.
Motor activity | up to 6 months
  Physical activity will be assessed using the Physical Activity Monitoring System (PAMsys).
Fatigue | up to 6 months
  Fatigue will be assessed using the Parkinson Fatigue Scale (PFS).
Strength | up to 6 months
  This will be assessed functionally using the 30 second Sit-To-Stand Test (30STS) for muscle strength.
Cognition | up to 6 months
  Cognition will be assessed using the Montreal Cognitive Assessment (MoCA).
Quality of life | up to 6 months
  This will be assessed by using a measure of disease-specific quality of life (Parkinson's Disease Questionnaire-39 (PDQ39)).
Long term behavioral change | up to 6 months
  All participants will track their participation in exercise and physical activity using an exercise diary for 6 months following the boot camp. Participants will be called monthly to reinforce completion of the exercise diary.
mini-Balance Evaluation Systems Test (mini-BESTest) | up to 6 months
  Performance-based balance tasks.
Falls self-efficacy | up to 6 months
  Activities Specific Balance Confidence Scale (ABC)
Fall Efficacy | Up to 6 months
  Self-report measurement tool: Falls Efficacy Scale (FES)
Fall catastrophization | Up to 6 months
  Self-report of fall catastrophization: Catastrophization about Falls Questionnaire (CAFS)
Physical activity | Up to 6 months
  Self-report measure physical activity: International Physical Activity Questionnaire (IPAQ)
Motor symptoms | Up to 6 months
  Unified Parkinson's Disease Rating Scale motor subscale (UDPRS III)
Fear of falling | Up to 6 months
  Self-report scale of avoidance behavior due to a fear of falling: Fear of Falls Avoidance Behavior Questionnaire (FFABQ)
Endurance | Up to 6 months
  Endurance will be assessed using the 6 Minute Walk Test (6MWT).
bone health | up to 6 months
  Bone health will be measured using bone mineral densiometry (BMD).
Mood | up to 6 months
  Mood will be measured using the Beck Depression Inventory.
Catalase | Up to 6 months
  Catalase concentrations from blood will be quantified utilizing enzyme-linked immunosorbent assays.
Cytokines | Up to 6 months
  Cytokine (TNFα, IL-6, IL-10) concentrations from blood will be quantified utilizing enzyme-linked immunosorbent assays.

OTHER OUTCOMES:
BDNF | up to 6 months
  Circulating BDNF concentrations from blood will be quantified utilizing enzyme-linked immunosorbent assays.

CONTACTS AND LOCATIONS:
Overall Officials: Merrill Landers, PT, DPT, PhD, Principal Investigator — UNLV
Locations (1):
- University of Nevada, Las Vegas, Las Vegas, Nevada, United States